CLINICAL TRIAL: NCT05955443
Title: iToBoS Prospective Data Acquisition Study
Brief Title: iToBoS Prospective Data Acquisition and Feasibility Study (Barcelona)
Acronym: iToBoS BCN
Status: Recruiting | Type: Observational
Sponsor: The University of Queensland (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Clare Primiero, Associate Investigator, The University of Queensland
Other Study IDs: BARCELONA_ITOBOS; 965221 (Other Grant/Funding Number: EU Horizon 2020)
Record Dates: First submitted 2023-06-28; First posted 2023-07-21 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Skin Cancer
Keywords: melanoma; skin examination; artificial intelligence; total body photography
MeSH Terms: conditions — Skin Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will be asked to provide a saliva or blood sample for genetic analysis. Some participants will already have a genetic sample with the hospital. In this case we will ask participant consent to access their biosample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is recruiting patients at their regular skin examination appointments to participate in research. Participation involves having 3D total body photography, completing a 10-15 minute questionnaire, and providing a genetic sample. Normally, the total body photography is part of the patients standard care, as is the collection of a genetic sample. Consenting to this study involves consenting to the use of total body photography images (de-identified), questionnaire answers, and genetic risk information to be used for developing AI algorithms for image analysis of skin lesions, and melanoma-risk profiling for patients.

DETAILED DESCRIPTION:
Patients are invited to participate at their regular skin examination visits at Hospital Clinic Barcelona. A member of the research team will read through the Participant Information and Consent Form (PICF) with the patient and answer any questions they may have. Once consent is given, the following study activities will take place.

1. Total Body Photography: this is done with the VECTRA machine that will require you to be photographed in your underwear. The VECTRA is a framework of 92 cameras which will simultaneously capture images of a patient holding one anatomical pose. VECTRA computer software is then used to construct a 3D avatar of the patient, enabling the image record of skin naevi. This imaging is normally part of the patient's skin examination visit. The images used for annotation in research will be de-identified (anonynmised) by firstly removing any images of the face and other identifying features (e.g. tattoos, scars, nipples), then processing the 3D avatar into small 2D images of 5x8cm section of skin. These methods are designed to protect patient privacy of images used for AI development.
2. Complete a Questionnaire: consists of 45 items/questions, taking approximately 10 minutes to complete. Questionnaire data is designed to collect information relevant to melanoma risk, while maintaining a low risk of being individually identifiable. topics cover include demographics, skin cancer history, sun/health behaviour, and phenotype information (e.g. hair/skin/eye colour).
3. Genetic sample: in some cases the hospital will already hold a genetic sample, in this case we ask patient consent to access this information. When no sample is on record, we will ask the patient to provide a saliva or blood sample for genetic analysis. Genetic information will be analysed by looking for single nucleotide polymorphisms (SNPs) relating to melanoma risk (approximately 80-100 SNPs to be analysed). A polygenic risk score (PRS) is then calculated based on the presence or absence of relevant SNPs. The final PRS will be used in the study (no individual genetic information will be shared outside the hospital.

All de-identified data (image, survey, and PRS) are then used by the iToBoS consortium to develop a cognitive assistant (AI model) to provide clinician support in screening for melanoma using total body photography.

ELIGIBILITY:
Inclusion Criteria:

* Over 18
* Able to provide informed consent

Exclusion Criteria:

* Unable to stand and hold anatomica pose for 3D total body photography

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are attending the Hospital Clinic de Barcelona for a standard skin examination will be approached to participate in the study. All participants will be adults, aged 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of skin diagnostic categories | Through study completion, an average of 1 year
  Images will be used to label different skin diagnostic categories. These labelled images are then used as a training dataset for machine learning in developing algorithms for skin lesion diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Malvehy, MD, Principal Investigator — Foundation Clinic for Biomedical Research
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided